CLINICAL TRIAL: NCT03033212
Title: Single-Level TLIF: Post-Fusion Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Research Manger, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MORPFR001
Record Dates: First submitted 2016-12-15; First posted 2017-01-26 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Degenerative Spinal Cord Disease
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Structured Rehabilitation (Experimental): Patients will begin Therapist-Guided Rehabilitation at 7 weeks postoperatively with a certified physical therapy. The patients will perform rehabilitation for 10 total weeks.
  Interventions: Other: Therapist-Guided Rehabilitation
- Delayed Rehabilitation (Experimental): Patients will begin Therapist-Guided Rehabilitation at 13 weeks postoperatively with a certified physical therapy. The patients will perform rehabilitation for 10 total weeks.
  Interventions: Other: Therapist-Guided Rehabilitation
- Self Rehabilitation (Active Comparator): Patients will begin Self-Guided Rehabilitation at 7 weeks postoperatively in a self-guided fashion. They will be provided with instructions for recommended exercises. They will undergo rehabilitation for a total of 10 weeks.
  Interventions: Other: Self-Guided Rehabilitation

INTERVENTIONS:
Other: Therapist-Guided Rehabilitation — Rehabilitation consists of exercises guided by a certified physical therapist. These exercises include: aerobics, walking tests, stability exercises, and strengthening exercises.
  Arms: Delayed Rehabilitation; Early Structured Rehabilitation
Other: Self-Guided Rehabilitation — Rehabilitation consists of self-guided exercises with provided instructions. These exercises include: aerobics, walking tests, stability exercises, and strengthening exercises.
  Arms: Self Rehabilitation

SUMMARY:
This investigation will assess how the timing and type of rehabilitation after a transforaminal lumbar interbody fusion will affect the efficacy of the surgical procedure. The efficacy of the procedure will be evaluated through patients' quality of life, measured by health-related quality of life questionnaires up to 24 months following the procedure. These measures will be compared to the patients' baseline value.

DETAILED DESCRIPTION:
Patients will undergo transforaminal lumbar interbody fusion for degenerative pathology at the L4-5 vertebral level. They will be randomized to one of three postoperative rehabilitation groups. Group 1 will receive "structured early rehabilitation" beginning at 7 weeks. Group 2 will receive "Delayed rehabilitation" beginning at 13 weeks postoperatively. Group 3 will undergo "Self Rehabilitation" beginning at 7 weeks postoperatively. Groups 1 and 2 will undergo rehabilitation under the supervision of a certified physical therapist for 10 total weeks. Group 3 will undergo non-supervised rehabilitation for 10 total weeks, and will be given educational materials regarding which exercises to perform and at which intervals.

ELIGIBILITY:
Inclusion Criteria:

i. Single-level L4-L5 TLIF for degenerative pathology, including: radiculopathy, neurogenic claudication, intervertebral disc disease, facet joint disease, degenerative spondylolisthesis, degenerative myelopathy degenerative kyphosis and scoliosis ii. Back and/or leg pain iii. Failed at least 3 months of conservative treatment

Exclusion Criteria:

i. Older than 65 years of age ii. Prior spinal surgery excluding laminectomy/discectomy iii. Greater than Grade 2 spondylolisthesis iv. Greater than 10 degrees scoliosis v. Not worked for greater than 6 months or unemployed as a result of lumbar condition vi. History of spinal infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index [ODI] Score at 2-years | Baseline, 2-year postoperative
  Oswestry Disability Index

SECONDARY OUTCOMES:
Radiographic fusion | Baseline, 1-year postoperative
  Radiographic fusion at L4-5 levels as measured by computed tomography scan
Change from baseline in walking ability at 2-years | Baseline, 2 years postoperative
  Walking test performed for 6 minutes
Change from baseline in walking speed at 2-years | Baseline, 2 years postoperative
  Walking test performed for 6 minutes
Change from baseline in Visual Analogue Scale [VAS] Pain Scores at 2-years | Baseline, 2 year postoperative
  Visual Analogue Scale
Change from baseline in Short-Form 12 [SF-12] Scores at 2-years | Baseline, 2 year postoperative
  Short-Form 12
Change from baseline PROMIS Physical Function Scores at 2-years | Baseline, 2 year postoperative
  PROMIS Physical Function
Change from baseline in Fear Avoidance Beliefs Metric at 2-years | Baseline, 2 year postoperative
  Fear Avoidance Beliefs Questionnaire
Change from baseline in Pain Catastrophization Metric at 2-years | Baseline, 2 year postoperative
  Pain Catastrophization Questionnaire
Change from baseline in Pain Neurophysiology Metric at 2-years | Baseline, 2 year postoperative
  Pain Neurophysiology Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Phillips, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Carla Edwards, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided